CLINICAL TRIAL: NCT05294705
Title: The Autism Biomarkers Consortium for Clinical Trials
Brief Title: The Autism Biomarkers Consortium for Clinical Trials: Confirmation Study
Acronym: ABC-CT CS
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Boston Children's Hospital (Other); Duke University (Other); Children's Hospital Los Angeles (Other); University of Washington (Other); Food and Drug Administration (FDA) (U.S. Federal Agency); University of Alabama at Birmingham (Other); University of California, Los Angeles (Other); Seattle Children's Hospital (Other); National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, James C. McPartland, Professor - Child Study Center, Yale University
Other Study IDs: 2000031989; U19MH108206 (NIH)
Record Dates: First submitted 2022-03-11; First posted 2022-03-24 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder
Keywords: Biomarkers
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Biospecimen Retention: Samples With DNA — Blood (DNA) samples will be collected from ASD participants and their biological parents at any timepoint after consent during this study. Briefly, blood samples can be collected by an appropriately trained research staff member, traveling phlebotomist, or at a clinic. A parent and a trained laboratory member may help alleviate any anxiety the child might have, including by the use of numbing cream or cooling spray as standard practice. Participants with ASD and their biological parent(s) will each have up to 30 mL of blood drawn. Blood draws for this study will be conducted in accordance with NIH guidelines. Study staff will share samples and study data via the NDAR and NIH/NIMH Data Repositories to create a community resource accessible for use by all qualified investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Autism Spectrum Disorder: During Screening Visits, the Autism Diagnostic Observational Schedule (ADOS) will be administered to confirm diagnosis. Criteria for group inclusion is: diagnosis of Autism Spectrum Disorder based on Diagnostic and Statistical Manual of Mental Disorders (DSM-5), the Autism Diagnostic Observation Schedule (ADOS-G), Brief Observation of Symptoms of Autism (BOSA), Childhood Autism Rating Scale-2(CARS-2) and the Autism Diagnostic Interview-Revised, short form (ADI-R). Diagnostic evaluations will be completed by research staff and supervised by a licensed psychologist.
- Typical Development: Typically Developing (TD) participants from each site will be roughly matched by age and sex to the ASD group.

SUMMARY:
This is a multicenter longitudinal study that aims to validate a set of measures that were previously identified as promising candidate biomarkers and/or sensitive and reliable objective measures of social function in ASD for potential use in clinical trials. The confirmation study will repeat the data collection and analysis protocols from the original ABC-CT study. This confirmation study will recruit 200 ASD and 200 TD comparison participants who are 6-11 years old, matching the overall sample size but providing a larger normative reference sample and greater statistical power for group comparisons.

DETAILED DESCRIPTION:
The goal of this consortium is to establish tools that can be used as biomarkers and/or sensitive and reliable objective assays of social function in autism spectrum disorder (ASD) clinical trials. Specifically, we aim to accelerate the development of effective treatments for social function in ASD by validating (a) outcome measures that will be sensitive and reliable assessments of response to treatment and (b) biomarkers in the domains of electroencephalography (EEG), eye-tracking (ET) and behavioral measures of social function to reduce heterogeneity of samples via stratification. The consortium will conduct a naturalistic, longitudinal study of school-aged (6-11 years) children with ASD and typical development (TD) with IQ ranging from 60-150 (ASD) and 80-150 (TD). Children will be assessed across three time points (T1: Baseline, T2: 6 weeks, T3: 24 weeks) using clinician and caregiver assessments along with a battery of conceptually related EEG and ET tasks and independent ratings of clinical status.

ELIGIBILITY:
Inclusion Criteria:

For All Subjects:

1. Males and Females Age 6 - 11 (less than 11 years and 6 months old at T1D1 unless all study procedures will be completed before the participant turns 12.0 and prior approval by the Principal Investigator is obtained).
2. Written parental permission, and child assents when applicable, obtained prior to any study procedures.
3. IQ 60-150 (ASD) and 80-150 (TD) as assessed by the Differential Ability Scales - 2nd Edition.
4. Participant and parent/guardian must be English speaking.

For ASD Participants (only):

1. Diagnosis of ASD based on Diagnostic and Statistical Manual of Mental Disorders (DSM-5), the Autism Diagnostic Observation Schedule (ADOS-2) or BOSA and the Autism Diagnostic Interview-Revised, short form (ADI-R). Diagnostic evaluations will be completed by research staff and supervised by a licensed psychologist.
2. If parents are biological, a minimum of the child and one parent will be required to consent to the blood draw procedure. It is preferred that the child and both biological parents participate in the blood draw procedure. The inability to obtain blood samples will not be exclusionary.

Exclusion Criteria:

For All Subjects:

1. Known genetic or neurological syndrome with an established link to autism (in addition to ASD for ASD participants)

   1. This does not include events in which the link to ASD is less well known/established (e.g., 16p11.2 CNVs, CHD8 mutations, Trisomy 21, 22q deletion syndrome, Dup 15q Syndrome).
   2. Specific cases will be discussed with the clinical team who will make a final determination, as needed.
2. History of epilepsy or seizure disorder

   a. This does not include history of simple febrile seizures or if the child is seizure free (regardless of the seizure type) for the past year.
3. Motor or sensory impairment that would interfere with the valid completion of study measures including significant hearing or vision impairment not correctable by a hearing aid or glasses/contact lenses. Children who wear bifocal or progressive lenses are not eligible.
4. Children who are taking neurological or psychiatric medications that are not stable on prescription or dose for 8 weeks prior to T1D1.

   a. Medication is not exclusionary. Children taking neurological or psychiatric medications, including anti epileptics and psychopharmacological agents, must be stable on the medication and dose for 8 weeks prior to T1D1.
5. History of significant prenatal/perinatal/birth injury as defined by birth <36 weeks AND weight <2000 grams (approximately 4.5.lbs).
6. History of neonatal brain damage. (e.g., with diagnosed hypoxic or ischemic event).
7. Any other factor that the investigator feels would make assessment or measurement performance invalid.
8. Participation in the original ABC-CT study.

For ASD Participants (only):

1. Any known environmental circumstance that is likely to account for autism in the proband.

For TD Participants (only):

1. Known historical diagnosis of ASD or a sibling with ASD.
2. Criteria score in the ASD range on the ADOS/BOSA at T1
3. Active psychiatric disorder (depression, anxiety, ADHD, etc.) and/or any current treatment (medication or other treatment) for a psychiatric condition.

   1. Participants will be screened using the Child/Adolescent Symptom Inventory (CASI- 5). Due to the instrument's high sensitivity and potential for false positives, any score in the clinical range will be reviewed by research staff for determination of eligibility.

Ages: 6 Years to 11 Years | Sex: All
Age Groups: Child
Study Population: 200 children with an autism spectrum disorder (ASD) between 6-11 years old, and 200 typically developing children between 6-11 years old
Sampling Method: Non-Probability Sample
Enrollment: 565 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
N170 Latency to Upright Human Faces | Baseline
  The N170 Latency to Upright Human Faces (N170 latency) is a scalp recorded EEG event-related potential (ERP) component elicited by perception of the upright human face. Recorded over the posterior-temporal right hemisphere, the latency (or speed) of the peak of the N170 ERP component occurs at approximately 200 msec in children aged 6 to 11 years of age.
Oculomotor Index of Gaze to Human Faces (OMI) | Baseline
  Onscreen gaze position data, reflected in percentage of foveation (angling of the eyes to focus on a particular object) to human faces (Face%) relative to total valid foveation time across three assays.
VABS: Vineland Adaptive Behavior Scales- III Socialization | Baseline
  Administered in person visit or via parent phone interview. The Socialization score is based on 3 subdomains of Interpersonal Relationships, Play & Leisure, Coping Scales. The V-Scaled scores, which are specifically designed to measure change over time, are only available for the subdomains. The primary norm-referenced scores for the subdomains are v-scale scores, which have a mean of 15 and standard deviation (SD) of 3. The Vineland-3 is a standardized measure of adaptive behavior--the things that people do to function in their everyday lives.
N170 Latency to Upright Human Faces | 6 weeks
  The N170 Latency to Upright Human Faces (N170 latency) is a scalp recorded EEG event-related potential (ERP) component elicited by perception of the upright human face. Recorded over the posterior-temporal right hemisphere, the latency (or speed) of the peak of the N170 ERP component occurs at approximately 200 msec in children aged 6 to 11 years of age.
Oculomotor Index of Gaze to Human Faces (OMI) | 6 weeks
  Onscreen gaze position data, reflected in percentage of foveation (angling of the eyes to focus on a particular object) to human faces (Face%) relative to total valid foveation time across three assays.
VABS: Vineland Adaptive Behavior Scales- III Socialization | 6 weeks
  Administered in person visit or via parent phone interview. The Socialization score is based on 3 subdomains of Interpersonal Relationships, Play & Leisure, Coping Scales. The V-Scaled scores, which are specifically designed to measure change over time, are only available for the subdomains. The primary norm-referenced scores for the subdomains are v-scale scores, which have a mean of 15 and standard deviation (SD) of 3. The Vineland-3 is a standardized measure of adaptive behavior--the things that people do to function in their everyday lives.
N170 Latency to Upright Human Faces | 24 weeks
  The N170 Latency to Upright Human Faces (N170 latency) is a scalp recorded EEG event-related potential (ERP) component elicited by perception of the upright human face. Recorded over the posterior-temporal right hemisphere, the latency (or speed) of the peak of the N170 ERP component occurs at approximately 200 msec in children aged 6 to 11 years of age.
Oculomotor Index of Gaze to Human Faces (OMI) | 24 weeks
  Onscreen gaze position data, reflected in percentage of foveation (angling of the eyes to focus on a particular object) to human faces (Face%) relative to total valid foveation time across three assays.
VABS: Vineland Adaptive Behavior Scales- III Socialization | 24 weeks
  Administered in person visit or via parent phone interview. The Socialization score is based on 3 subdomains of Interpersonal Relationships, Play & Leisure, Coping Scales. The V-Scaled scores, which are specifically designed to measure change over time, are only available for the subdomains. The primary norm-referenced scores for the subdomains are v-scale scores, which have a mean of 15 and standard deviation (SD) of 3. The Vineland-3 is a standardized measure of adaptive behavior--the things that people do to function in their everyday lives.

SECONDARY OUTCOMES:
Aberrant Behavior Checklist (ABC) | Baseline, 6 weeks and 24 weeks
  The Aberrant Behavior Checklist (ABC) is a symptom checklist for assessing problem behaviors of children and adults with neurodevelopmetnal disorder at home, in residential facilities, ICFs/MR, and work training centers. It is also useful for classifying problem behaviors of children and adolescents with neurodevelopmetnal disorder in educational settings, residential and community-based facilities, and developmental centers.
Autism Impact Measure (AIM) | Baseline, 6 weeks and 24 weeks
  The Autism Impact Measure (AIM) uses a 2-week recall period with items rated on two corresponding 5-point scales (frequency and impact)
Behavior Assessment System for Children -3 (BASC-3) | Baseline
  The Behavior Assessment System for Children, Third Edition (BASC-3) offers several different forms designed to aid in collecting information regarding at-risk adaptive behavioral and/or emotional problems.
Child and Adolescent Symptom Inventory 5 (CASI-5) | Baseline and 24 weeks
  The Child & Adolescent Symptom Inventory-5 (CASI-5) is a behavior rating scale for DSM-5-defined emotional and behavioral disorders in youths between 5 and 18 years old.
PDD Behavior Inventory (PDD-BI) | Baseline, 6 weeks and 24 weeks
  The PDD-BI is an assessment tool for children on the autism spectrum. PDDBI profiles can provide guidance to clinicians regarding the child's problems as perceived by the informants, how a particular child compares to most children their age with ASD, and the skills and abilities of the child.
Social Responsiveness Scale 2 (SRS-2) | The Social Responsiveness Scale 2 (SRS-2) is completed in just 15 to 20 minutes and identifies social impairment associated with autism spectrum disorders (ASDs) and quantifies its severity.
  Baseline and 24 weeks
Cognitive Assessment | Differential Ability Scales - Second Edition; DAS-II (Elliott C, 2007): The DAS-II is a clinical instrument designed to assess cognitive ability include variables such as verbal cluster, spatial cluster, nonverbal cluster, special nonverbal composite and
  Baseline and 24 weeks
Resting State EEG | Baseline, 6 weeks and 24 weeks
  Resting State EEG (Eyes Open) provides a reference for the event-related EEG measures and a baseline biomarker of EEG spectral power across frequencies, neurofunctional connectivity and coherence, and hemispheric asymmetry and will always be done prior to the other EEG paradigms. Participants will be presented with non-social, abstract moving videos in random order.
Faces Processing EEG | Faces processing is a foundation for social perception and attention and serves as a promising and robust biomarker of social impairment in ASD and a potential index of subgroup differences. As the primary non-resting paradigm, the FACES task will always
  Baseline, 6 weeks and 24 weeks
Visual Evoked Potentials (VEPs) EEG | Baseline, 6 weeks and 24 weeks
  Visual Evoked Potentials (VEPs) index low-level visual processing and reflect the functional integrity of the visual pathway. VEPs reflect excitatory (glutamatergic) and inhibitory (GABAergic) activity and may index subgroups of ASD with low-level visual impairments. VEPs also serve as a control for assessment of higher-order activity in social visual paradigms. Subjects will be presented with black and white checkerboards that reverse phase at a defined interval. The order of the VEP and Biomotion paradigms will be counterbalanced.
Eye-Tracking (ET) Activity Monitoring Task | Baseline, 6 weeks and 24 weeks
  ET Paradigms will be administered in counterbalanced blocks, one on each day of each screening or study visits. Both blocks will include all the tasks but in different orders. The length of individual paradigms ranges from 1 to 8.5 mins.
  Activity Monitoring Task is measured following central fixation. Children will be presented with multiple activity monitoring trails depicting two actresses engaging in a controlled joint activity such as assembling a puzzle.
Eye-tracking (ET) Interactive Social Task (IST) | Baseline, 6 weeks and 24 weeks
  ET Paradigms will be administered in counterbalanced blocks, one on each day of each screening or study visits. Both blocks will include all the tasks but in different orders. The length of individual paradigms ranges from 1 to 8.5 mins.
  Interactive Social Task (IST) is taps similar constructs as the activity monitoring task in a more naturalistic, dynamic, and complex context. Following a central fixation, children will be presented with interactive social trails in which two children engage in a natural interactive play session.
Eye-tracking (ET) Pupillary Light Reflex Task | Baseline, 6 weeks and 24 weeks
  ET Paradigms will be administered in counterbalanced blocks, one on each day of each screening or study visits. Both blocks will include all the tasks but in different orders. The length of individual paradigms ranges from 1 to 8.5 mins.
  Pupillary Light Reflex (PLR) Task is measured following a stimuli that consist of a central fixation point on a black background that flashes white for 133 milliseconds. The constriction of the pupil in response to a bright flash indexes function of the parasympathetic nervous system.
Eye-tracking (ET) Static Social Scenes Task | Baseline, 6 weeks and 24 weeks
  ET Paradigms will be administered in counterbalanced blocks, one on each day of each screening or study visits. Both blocks will include all the tasks but in different orders. The length of individual paradigms ranges from 1 to 8.5 mins. Color images depicting 12 different female faces with direct gaze and the same faces with averted gaze will be presented. Twelve different exemplars from each of five categories (alarm clocks, mobile phones, birds, cars, and shoes) will be used as distracters. Twelve different slides will each contain six images (one face and five distracters, one from each category) placed at an equal distance from the center of the screen. Each slide contains a different set of six images, each image being shown only once in the experiment. This measure examines scanning patterns towards arrays of objects, synthetic stimuli, and faces as well as towards more complex naturalistic (static) scenes. This task examines complex scene processing and attentional selection.
NEPSY-II | Baseline, 6 weeks and 24 weeks
  NEPSY-II - Memory for Faces Subtest (administered to all ages): The NEPSY-II Memory for Faces subtest entails viewing a series of faces and having the child identify the sex of each face. The child is then shown three faces at a time and required to identify the previously seen face.

CONTACTS AND LOCATIONS:
Overall Officials: James McPartland, PhD, Principal Investigator — Yale University
Locations (5):
- United States (5):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Yale Child Study Center, New Haven, Connecticut
  - Boston Children's Hospital, Boston, Massachusetts
  - Duke, Durham, North Carolina
  - Unviersity of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
IPD will be uploaded to the National Institute of Mental Health Data Archeive.
Time Frame: Data is uploaded every 6 months throughout the study.
Access Criteria: Per NDA access requirements.
URL: https://nda.nih.gov/